CLINICAL TRIAL: NCT00003028
Title: Phase I Study to Determine the Safety of MEN-10755 (BMS-195615) in Patients With a Solid Tumor on a Short I.V. Infusion Given Once Every 3 Weeks
Brief Title: MEN-10755 in Treating Adults With Recurrent or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16969; EORTC-16969
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — sabarubicin

INTERVENTIONS:
Drug: sabarubicin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of MEN-10755 in treating adults who have recurrent or refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD) of MEN-10755 in patients with recurrent or refractory adult solid tumors. II. Determine the qualitative and quantitative toxic effects of MEN-10755 and study the predictability, duration, intensity, onset, reversibility, and dose relationship of the toxic effects in these patients. III. Propose a safe dose for phase II study. IV. Assess the pharmacokinetics of MEN-10755 at different dose levels in these patients. V. Document any possible antitumor activity of MEN-10755.

OUTLINE: This is an open label, nonrandomized study. Patients receive MEN-10755 as a single 15 minute intravenous infusion every 3 weeks, or upon recovery from toxicity. Doses will be escalated in decreasing rates and depending on the clinical judgement of the investigator. The MTD is the dose at which dose limiting toxicity is observed in at least 2 of 6 patients at a given dose level. Patients will be removed from the study if cardiac toxicity, disease progression, or renal, cardiac or pulmonary decline is present.

PROJECTED ACCRUAL: At least 5 evaluable patients will be enrolled.

ELIGIBILITY:
DISEASE CHARACTERISTICS: See General Eligibility Criteria

PATIENT CHARACTERISTICS: Age: 18 and over Performance Status: WHO 0-2 Life Expectancy: At least 3 months Hematopoietic: ANC at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Liver function tests no greater than 2 times upper limit of normal (ULN) (unless related to liver metastases, then no greater than 5 times ULN) Renal: Creatinine no greater than 1.4 mg/dL Creatinine clearance at least 60 mL/min Cardiovascular: LVEF greater than 50% (measured by MUGA scan) Other: Not pregnant or nursing Effective contraceptive method must be used during study No active bacterial infections No other nonmaliganant diseases No history of alcoholism or drug abuse No psychosis

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy within 4 weeks of study Concurrent use of growth factors is allowed in cases of febrile neutropenia (prophylactic use not allowed) Chemotherapy: No prior chemotherapy within 4 weeks of study No prior nitrosoureas, mitomycin, or high dose carboplatin within 6 weeks of study Endocrine therapy: No concurrent corticosteroids (unless approved by clinical investigator) Radiotherapy: No prior radiotherapy within 4 weeks of study No prior extensive radiotherapy within 6 weeks of study Surgery: Not specified Other: No prior experimental therapy No prior anthracyclines or anthracenediones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 1997-04

CONTACTS AND LOCATIONS:
Overall Officials: Per Dombernowsky, MD, Study Chair — Copenhagen County Herlev University Hospital
Locations (49):
- Ludwig Boltzmann - Institute for Applied Cancer Research, Vienna, Austria
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Herlev Hospital - University Hospital of Copenhagen, Herlev
- France (14):
  - Institut Bergonie, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lute Contre le Cancer,Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - CHU de la Timone, Marseille
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Institut Curie - Section Medicale, Paris
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Hopital Paul Brousse, Villejuif
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Martin Luther Universitaet, Halle
  - Universitats-Krankenhaus Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Nurnberg, Nuremberg (Nurnberg)
- University of Ioannina, Ioannina, Greece
- Israel (2):
  - Rambam Medical Center, Haifa
  - Schneider Children's Medical Center of Israel, Petah Tikva
- Italy (5):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Istituto Europeo Di Oncologia, Milan
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
  - San Raffaele Hospital, Rome
  - Istituti Fisioterapici Ospitalieri - Roma, Rome
- Netherlands (5):
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Ziekenhuis der Vrije Universiteit, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - University Medical Center Nijmegen, Nijmegen
  - Rotterdam Cancer Institute, Rotterdam
- Norwegian Radium Hospital, Oslo, Norway
- Instituto Portugues de Oncologia de Francisco Gentil, Lisbon, Portugal
- Hospital Universitario 12 de Octubre, Madrid, Spain
- Switzerland (5):
  - University Hospital, Basel
  - Ospedale San Giovanni, Bellinzona
  - Inselspital, Bern, Bern
  - Clinique De Genolier, Genolier
  - Kantonsspital - Saint Gallen, Sankt Gallen
- United Kingdom (4):
  - Royal Marsden NHS Trust, London, England
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Western General Hospital, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland